CLINICAL TRIAL: NCT05161078
Title: Improving Continuous Renal Replacement Therapy (CCRT) Outcomes in Neonates and Infants Through Interdisciplinary Collaboration
Brief Title: Improving Continuous Renal Replacement Therapy Outcomes in Neonates and Infants Through Interdisciplinary Collaboration
Acronym: ICONIIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Mozarc Medical US LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ICONIIC
Record Dates: First submitted 2021-11-23; First posted 2021-12-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury; Chronic Kidney Diseases; Renal Dialysis
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples Without DNA — Urine will be collected via natural void or collected in some other manner if ordered per standard of care. Blood specimen will be obtained from residual clinical specimen only. All specimen will be stored for future unspecified research at Cincinnati Children's.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Patients Enrolled: Patients will be treated with CARPEDIEM per standard of care.
  Interventions: Device: CARPEDIEM

INTERVENTIONS:
Device: CARPEDIEM — CARPEDIEM treatment as per local standard of care

SUMMARY:
To date, little knowledge exists related to the use of hemodialysis (HD) in infants and has been limited to mainly single center studies. The CARPEDIEM (CArdio-Renal PEdiatric Dialysis Emergency Machine) device, which can be used to provide hemodialysis in infants, has been launched in the United States. This study/registry is designed to obtain data on critically ill infants who require HD using the CARPEDIEM device to understand the indications for initiation, best practice in prescribing and performing treatment, expected treatment course, and outcomes of a dedicated infant continuous renal replacement therapy (CRRT) machine.

DETAILED DESCRIPTION:
This is a retrospective and prospective, multicenter observational quality improvement study and research registry. Infants undergoing renal replacement therapy utilizing CARPEDIEM for hemodialysis will be enrolled in the study for observation. There are two arms to this study, one for quality improvement and one for research purposes. Patients enrolled in this study have the option to participate additionally in either biospecimen collection, long term follow up after CARPEDIEM, or both. Urine specimen will be collected from fresh voids, but all blood specimen will be obtained from residual clinical specimen. Investigators hope to gain more information into use, treatment course, and outcomes from infants requiring treatment with the CARPEDIEM device.

ELIGIBILITY:
Inclusion Criteria:

* Treated with CARPEDIEM as part of standard of care at a participating institution within the United States

Exclusion Criteria:

* Parents/legally authorized representative unable or unwilling to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with CARPEDIEM as part of standard of care at a participating institution's Neonatal Intensive Care Unit (NICU), Cardiac Intensive Care Unit (CICU), or Pediatric Intensive Care Unit (PICU).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of CARPEDIEM filters to meet prescribed treatment length | 24 hours
  Comparing actual time of treatment of each CARPEDIEM filter to the initial prescribed length of treatment at the time of filter initiation
Rate of patient survival | through hospital discharge, an average of less than 1 year
  Percent of patients treated with the CARPEDIEM who survive to hospital discharge
Rate of renal recovery | through hospital discharge, an average of less than 1 year
  Excluding patients with End Stage Renal Disease (ESRD), percent of patients treated with the CARPEDIEM who recover baseline renal function as measured by liberation from dialysis and serum creatinine returning to within less than a 50% increase over baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Slagle, MD, Principal Investigator — Cincinnati Children's
Locations (9):
- United States (9):
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided